CLINICAL TRIAL: NCT04757753
Title: Evaluation of the Efficacy Rate of Endodontic Treatment at 2 Years After Root Canal Filling With a Ready-to-use Root Canal Sealer PA1704 Versus BioRoot™ RCS: a Randomized Controlled Trial
Brief Title: Root Canal Obturation With a Ready-to-use Root Canal Sealer (PA1704) Versus BioRoot™ RCS: a Randomized Controlled Trial
Acronym: OPTIFILL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Septodont (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20/001; 2020-A01790-39-PP (Other: French National Agency of Medicines and Health products); CIV-BE-20-10-034945 (Other: Belgium Federal Agency for Medicines and Health products)
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Root Canal Obturation
Keywords: endodontic treatment; root canal sealer; periapical lesion

STUDY DESIGN:
Intervention Model Description: Study subject (tooth) will be randomized in a 1:1 allocation ratio between the 2 treatment groups; the allocation will be stratified by the endodontic indication, i.e. primary or secondary root canal treatment, to enhance balance.
Who Masked: Outcomes Assessor
Masking Description: Blinding will be done to the assessors who analyzed radiographs to reduce bias to healing assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ready-to-use root canal sealer: PA1704 (Experimental): PA1704 is used in combination with gutta percha points for the permanent obturation of root canals.
  Interventions: Device: ready-to-use root canal sealer: PA1704
- root canal sealer: BioRoot™ RCS (Other): BioRoot™ RCS is used in combination with gutta percha points for the permanent obturation of root canals.
  Interventions: Device: root canal sealer: BioRoot™ RCS

INTERVENTIONS:
Device: ready-to-use root canal sealer: PA1704 — The participant will be treated with the ready-to-use root canal sealer (PA1704) in combination with gutta percha.
  Arms: ready-to-use root canal sealer: PA1704
Device: root canal sealer: BioRoot™ RCS — The participant will be treated with BioRoot™ RCS sealer in combination with gutta percha.
  Arms: root canal sealer: BioRoot™ RCS

SUMMARY:
The study design is a multicentric randomized controlled non-inferiority trial. 160 subjects (teeth) requiring a primary or a secondary root canal treatment will be enrolled in 2 groups (80 in each group). The aim of the study is to assess the efficacy rate and the safety 2 years after root canal obturation undertaken using a ready-to-use calcium silicate sealer (PA1704) compared to the control calcium silicate sealer BioRoot™ RCS.

Procedures of root canal treatment will be conventional and standardized for all investigational centers. The canals will be cleaned, shaped and then obturated using a calcium silicate sealer (the ready to use sealer PA1704 or BioRoot™ RCS) with a single cone technique or cold lateral condensation of gutta-percha. Follow-up assessments will be conducted at 6, 12 and 24 months in both groups. The performance and safety of the sealer PA1704 will also be evaluated at 3.5 and 5 years after surgery. Retroalveolar radiographs will be taken at each study visit. The preoperative, postoperative and follow-up clinical and radiographic data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (age ≥ 18 years)
* Patient requiring a primary or a secondary root canal obturation on a single or multi-rooted tooth,
* Patient geographically stable who can be followed by the same investigator site for 2 years,
* Informed consent signed,
* Patient with social protection

Exclusion Criteria:

* Patient with one or more documented contraindication to endodontic treatment,
* Contraindication to the use of calcium silicate root canal sealer, such as an immature tooth or a known hypersensitivity to one component of the sealer formula,
* Endodontic treatment on tooth with calcified root canal assessed radiographically,
* Endodontic treatment on tooth with suspected perforation,
* Patient with an uncontrolled systemic disease such as diabetes or thyroid disorders, or with an immunocompromised condition or who has undergone radiation therapy to the jaw.
* Patient suffering from uncontrolled active periodontitis, not supported
* Participation to another interventional clinical study at the same time,
* Vulnerable subjects referred to in articles L.1121-5 to 8 and L.1122-1-2 of the Public Health Code and article 66 of Regulation (EU) 2017/745 on medical devices are excluded from the investigation (such as known pregnancy or lactation, patients with legal protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Simon, Pr, DDS, Principal Investigator — Cabinet dentaire Jeanne d'Arc - ROUEN (76000) - France
Locations (5):
- Cliniques Universitaires Saint-Luc, Département de Médecine Dentaire et de Stomatologie, Brussels, Belgium
- France (4):
  - Centre de santé dentaire Flandre, Paris
  - Cabinet dentaire, Rennes
  - Cabinet dentaire Jeanne d'Arc, Rouen
  - Cabinet dentaire, Saint-Grégoire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Simon S, Beauquis J, Colombel H, Dorn A, Marchi V, Robert S, Souleau G, Ravalec N, Huguet-Jaime F, Chazaud K, Serandour AL, Ournid N, Leprince JG. Clinical efficacy of root canal treatment at 2 years using a new ready-to-use injectable calcium silicate-based sealer: A multicentric randomised controlled trial. Int Endod J. 2025 Sep;58(9):1420-1432. doi: 10.1111/iej.14265. Epub 2025 Jun 10. PMID 40491343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical investigation OPTIFILL has been conducted in a total of 7 investigational sites: 6 centers were in France and 1 center was in Belgium. Investigators are dental surgeons (endodontists or general dentists) from private practice offices or hospital.
  Recruitment was conducted over 9 months, between November 2020 and July 2021.
Pre-assignment Details: No randomization in case of screen failure or eligibility criteria noncompliance.
Groups:
- PA1704: As a ready-to-use root canal sealer, PA1704 is used in combination with gutta percha points for the permanent obturation of root canals.
- BioRoot™ RCS: As a ready-to-use root canal sealer, BioRoot™ RCS is used in combination with gutta percha points for the permanent obturation of root canals.
Period: Overall Study
Arm/Group | PA1704 | BioRoot™ RCS
Started | 77 | 83
Completed | 66 | 71
Not Completed | 11 | 12
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Endodontic treatment failure | 1 | 2
Not completed — Tooth fracture/extraction | 3 | 0

BASELINE CHARACTERISTICS:
Population: All the randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | PA1704 | BioRoot™ RCS | Total
Number analyzed (Participants) | 77 | 83 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (16.1) | 46.3 (16.3) | 48.5 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 46 | 77
  Male | 46 | 37 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 11 | 13 | 24
  France | 66 | 70 | 136
Tooth type [Count of Participants; unit: Participants] — Description of teeth to be treated at baseline
  Participants
    Incisor | 8 | 2 | 10
    Canine | 3 | 5 | 8
    Premolar | 22 | 31 | 53
    Molar | 44 | 45 | 89
Number of canals to treat [Count of Participants; unit: Participants]
  1 canal | 23 | 22 | 45
  2 canals | 10 | 16 | 26
  3 canals | 26 | 24 | 50
  4 canals | 17 | 20 | 37
  5 canals | 1 | 1 | 2
Type of endodontic treatment [Count of Participants; unit: Participants]
  Initial treatment | 55 | 59 | 114
  Retreatment | 22 | 24 | 46
Pulp diagnosis among initial treatments [Count of Participants; unit: Participants] — Population: Information regarding the diagnosis of the tooth pulp is given for initial treatment subpopulation only, since there is no pulp anymore in the retreatment subpopulation.
  Participants
    number analyzed (Participants) | 55 | 59 | 114
    Irreversible pulpitis | 14 | 11 | 25
    Necrotic pulp | 28 | 31 | 59
    Live pulp with endodontic treatment indication | 13 | 17 | 30
Apical lesion [Count of Participants; unit: Participants] — Number of patients with an apical lesion before the treatment
  Participants | 34 | 35 | 69
Symptomatic tooth [Count of Participants; unit: Participants] — Number of patients with a symptomatic tooth before the treatment
  Participants | 28 | 32 | 60

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Rate of Root Canal Obturation
Description: Efficacy rate of root canal obturation using clinical and radiological criteria.
  A successfull treatment is defined in this study, based on some loose criteria, as: a functional tooth with no lesion on the radio, or a functional tooth with a size reduction of the lesion on the radio, or a functional tooth with a lesion size stabilisation.
Time Frame: 24 months post-treatment
Population: Per Protocol population: All patients for whom the efficacy rate of root canal obturation is measurable at 24 months post-treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PA1704 | BioRoot™ RCS
Number analyzed (Participants) | 67 | 73
Participants
  Successfull treatment | 61 | 66
  Unsuccessfull treatment | 6 | 7
Statistical Analysis 1: Comparison: PA1704 vs BioRoot™ RCS; The statistical analysis was done on the proportion difference of the treatment efficacy, defined on loose criteria, at 24 months, in PP population; Test type: Non-Inferiority — πN = 2-year successful treatment rate of PA1704 πR = 2-year successful treatment rate of BioRoot™ RCS Δ = πN - πR ΔL = non-inferiority margin fixed to 13% or 0.13 Hypotheses are : H0 : Δ ≤ -ΔL H1 : Δ > -ΔL The χ2 of Dunnett & Gent is used to assess the non-inferiority; p = 0.03, Chi-squared, Corrected — A priori threshold for statistical significance was < 0.05; Mean Difference (Final Values) = 0.006, 90% CI 2-sided [-0.0074 to 0.0087]

2. Secondary Outcome: Efficacy Rate of Root Canal Obturation
Description: Efficacy rate of root canal obturation using clinical and radiological criteria.
  A successfull treatment is defined in this study, based on some loose criteria, as: a functional tooth with no lesion on the radio, or a functional tooth with a size reduction of the lesion on the radio, or a functional tooth with a lesion size stabilisation.
  The efficacy rates was compared between the 2 groups at 12-months post-treatment.
Time Frame: 12 months post-treatment
Population: mITT Population (12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | PA1704 | BioRoot™ RCS
Number analyzed (Participants) | 68 | 76
Participants
  Successful treatment | 63 | 69
  Unsuccessful treatment | 5 | 7

3. Secondary Outcome: Efficacy Rate of Root Canal Obturation
Description: Efficacy rate of root canal obturation using clinical and radiological criteria.
  A successfull treatment is defined in this study, based on some loose criteria, as: a functional tooth with no lesion on the radio, or a functional tooth with a size reduction of the lesion on the radio, or a functional tooth with a lesion size stabilisation.
  The efficacy rates was compared between the 2 groups at 6-months post-treatment.
Time Frame: 6 months post-treatment
Population: mITT Population (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | PA1704 | BioRoot™ RCS
Number analyzed (Participants) | 71 | 79
Participants
  Successfull Treatment | 68 | 75
  Unsuccessfull Treatment | 3 | 4

4. Secondary Outcome: Radiological Evaluation of the Canal Obturation
Description: Radiological evaluation of the level of apical obturation and density.
  The level of apical obturation and density is measured by the Investigators on the retroalveolar radios, like the "Sufficient radio-opacity" of the ready-to-use root canal sealer under investigation, "Presence of at least one bubble (void) in the filling material", and "If extruded material at T0, extruded material still presents in the periapical space".
Time Frame: 24-months post-treatment
Population: mITT population (24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | PA1704 | BioRoot™ RCS
Number analyzed (Participants) | 66 | 71
Participants
  Sufficient radio-opacity | 65 | 71
  Presence of at least one bubble (void) in the filling material | 2 | 5
  If extruded material at T0, extruded material still presents in the periapical space: number analyzed (Participants) | 31 | 21
  If extruded material at T0, extruded material still presents in the periapical space | 26 | 15

5. Secondary Outcome: Postoperative Pain
Description: The pain is assessed by patients in a diary using a Visual Analogue Scale (VAS: 0-100 mm, from no pain to max pain) at different times after endodontic treatment (at the end of the root canal obturation, 12h postoperative, 24h, Day 2, Day 3, Day 7). The maximum pain felt will be compared between the 2 groups.
  To note: the endodontic treatment was performed in 2 sessions for some patients. For those patients, there is an additional pain evaluation done before the session 2.
Time Frame: Before endodontic treatment*; before session#2 initiation**; T0 (after canal obturation); 12; 24; 48; & 72h; 7 days after endodontic treatment. *Evaluation on same day for 1-session treatment; up to 18 days before if 2 sessions needed. **On same day.
Population: ITT population
Measure: Mean (Standard Deviation); unit: millimeters on the VAS
Arm/Group | PA1704 | BioRoot™ RCS
Number analyzed (Participants) | 76 | 80
millimeters on the VAS
  Before endodontic treatment initiation: number analyzed (Participants) | 73 | 71
  Before endodontic treatment initiation | 6.0 (16.2) | 7.1 (15.3)
  Before session 2 initiation: number analyzed (Participants) | 7 | 8
  Before session 2 initiation | 1.9 (3.3) | 0.1 (0.4)
  Post-operative pain At T0 | 2.6 (5.8) | 3.6 (8.4)
  Post-operative pain At 12 hours: number analyzed (Participants) | 73 | 73
  Post-operative pain At 12 hours | 12.3 (17.5) | 11.6 (18.6)
  Post-operative pain At 24 hours: number analyzed (Participants) | 68 | 73
  Post-operative pain At 24 hours | 6.5 (11.9) | 8.8 (16.6)
  Post-operative pain At 48 hours: number analyzed (Participants) | 72 | 77
  Post-operative pain At 48 hours | 5.0 (10.4) | 7.1 (15.4)
  Post-operative pain At 72 hours: number analyzed (Participants) | 73 | 73
  Post-operative pain At 72 hours | 3.8 (11.3) | 2.9 (7.8)
  Post-operative pain At 7 days: number analyzed (Participants) | 62 | 64
  Post-operative pain At 7 days | 0.5 (1.1) | 0.7 (1.8)

6. Secondary Outcome: Use of Oral Pain Treatment
Description: Patients reported the consumption of analgesic treatment in a diary. The percentage of patients who took oral pain medication will be compared between the 2 groups.
Time Frame: From Day 0 to Day 7
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | PA1704 | BioRoot™ RCS
Number analyzed (Participants) | 77 | 83
Participants
  Patients who used an oral pain treatment between T0 and D7 | 37 | 39
  Reasons for using an oral pain treatment is a dental pain: number analyzed (Participants) | 37 | 39
  Reasons for using an oral pain treatment is a dental pain | 24 | 25
  Reasons for using an oral pain treatment is an other pain: number analyzed (Participants) | 37 | 39
  Reasons for using an oral pain treatment is an other pain | 11 | 12
  Reasons for using an oral pain treatment is both an oral and another pain: number analyzed (Participants) | 37 | 39
  Reasons for using an oral pain treatment is both an oral and another pain | 2 | 2

ADVERSE EVENTS:
Time Frame: 2 years post-treatment
Arm/Group | PA1704 | BioRoot™ RCS
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/83
Serious Adverse Events (participants affected / at risk) | 2/77 | 0/83
Other Adverse Events (participants affected / at risk) | 19/77 | 20/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA1704 (N=77) | BioRoot™ RCS (N=83)
Embolism pulmonary (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Embolism pulmonary, not related to the Investigational Medical Device
Spinal Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Surgery to treat a spinal hernia, not related to the investigational medical device
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA1704 (N=77) | BioRoot™ RCS (N=83)
Tooth fracture (General disorders) | 3 (3) | 3 (3)
Tooth extraction (General disorders) | 3 (3) | 3 (3)
Tooth pain (General disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 9 (9) | 7 (7)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Postoperative pain (General disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT04757753/Prot_SAP_000.pdf